CLINICAL TRIAL: NCT02886962
Title: Study of the Benefit / Risk Ratio of Oral Anticoagulation in Hemodialysis Patients With Atrial Fibrillation
Brief Title: Oral Anticoagulation in Haemodialysis Patients
Acronym: AVKDIAL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6396
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No anticoagulation (Experimental): No oral anticoagulation, and no monitoring of the INR.
  Interventions: Biological: No oral anticoagulation
- Oral anticoagulation with vitamin K antagonists (Active Comparator): VKA use as recommended in the guidelines with INR target range between 2 and 3. Daily administration or thrice weekly at the end of dialysis sessions upon Nephrologist's choice.
  Antiplatelet therapy will be provided only if recent acute coronary syndrome (< 6 months) or active coronary stent. Aspirin should be preferred in dialysis patients as clopidogrel has an unpredictable reduced activity and there is no safety data on combination of VKA with prasugrel or ticagrelor in this population.
  Interventions: Drug: Oral anticoagulation with vitamin K antagonists

INTERVENTIONS:
Biological: No oral anticoagulation — No oral anticoagulation, and no monitoring of the INR.
  Arms: No anticoagulation
Drug: Oral anticoagulation with vitamin K antagonists — Vitamin K antagonist prescription with INR target between 2 and 3 as recommended in the guidelines.
  Administration once daily or at the end of each dialysis session, according to the nephrologist choice.
  INR monitoring at least once per week
  Arms: Oral anticoagulation with vitamin K antagonists

SUMMARY:
Guidelines recommend oral anticoagulation with vitamin K antagonists for atrial fibrillation whenever the CHADS2VASC score is superior or equal to 2. As there are no specific guidelines for the hemodialysis patients with atrial fibrillation, the general guidelines apply. However, several retrospective studies suggest that these patients do not benefit from the oral anticoagulation regarding the risk of stroke and may even experience more bleedings and deaths.

The aim of this prospective study is to prospectively compare the hemorrhagic and thrombotic risks of oral anticoagulation in comparison with no anticoagulation in hemodialysis patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Patient on hemodialysis treatment for at least 1 month
* Patient with a history of, or presenting a new episode of atrial fibrillation (either permanent or paroxysmal).
* Patient with a CHADS2VASC score ≥2
* Patient with high risk of bleeding as defined by (1) HASBLED score ≥3 OR (2) HASBLED ≥ CHADS2VASC score, OR (3) recent history of severe bleeding (type 3a, 3b, 3c), particularly cerebral or gastrointestinal, OR (4) prior recurrent (>2) history of falls.
* Patient capable of understanding information about the study and of giving his/her consent
* Patient informed of the preliminary medical exam results
* Patient with healthcare insurance
* Written consent signed

Exclusion Criteria:

* Formal indication to oral anticoagulation beside atrial fibrillation (mechanic heart valves, recurrent thrombophlebitis, antiphospholipid syndrome)
* Life expectancy < 6 months (e.g., terminal cancer)
* Live donor transplantation scheduled within 6 months
* Pregnancy (β-HCG blood-based assay)or nursing (lactating) women
* Women of child bearing potential, unless they are using an effective method of birth control
* Patient under legal guardianship
* Patients under law protection
* Known hypersensibility to coumadin or indoine derivatives or to any excipients (CI to oral AVK)
* Severe liver failure (CI to oral AVK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of severe bleedings and thrombosis of oral anticoagulation versus no anticoagulation in hemodialysis patients with atrial fibrillation | 2 years

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - Service de Néphrologie et médecine interne, Amiens
  - CHRU d'Angers - Service de Néphrologie, Angers
  - Service Néphrologie, Dialyse, Transplantation, Caen
  - Pathologie Rénale, Chambéry
  - Service de Néphrologie, Cherbourg-Octeville
  - Aural Colmar, Colmar
  - Service de néphrologie, Colmar
  - Service de néphrologie, Dijon
  - Aurad Aquitaine, Gradignan
  - Centre Hospitalier de Haguenau - service de Néphrologie, Haguenau
  - AURAL Haguenau, Haguenau
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Clinique Bouchard, Marseille
  - Service de Néphrologie, Nancy
  - ECHO de Nantes, Nantes
  - Service de Néphrologie, Nantes
  - AURA Paris Plaisance, Paris
  - Hôpital Tenon - Service de Néphrologie, Paris
  - Service de néphrologie, Rennes
  - ECHO CA Laennec, Saint-Herblain
  - NéphroCare Tassin-Charcot, Sainte-Foy-lès-Lyon
  - AURAL st Anne, Strasbourg
  - Service de Néphrologie, Strasbourg
  - Centre Hospitalier Bretagne-Atlantique, Vannes
  - Calydial CH Lucien Hussel, Vienne

IPD SHARING:
Plan to Share IPD: No